CLINICAL TRIAL: NCT03263234
Title: Circadian Adjusted LED Light's Effect on Sleep, Circadian Rhythm, and Well-being in People Living in Elderly Housing: a Cross-over Non-blinded Randomized Trial.
Brief Title: Circadian Adjusted LED Light's Effect in People Living in Elderly Housing
Acronym: Lightel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ove Andersen (Other)
Collaborators: Chromaviso A/S (Other); Albertslund Kommune (Unknown); Aalborg University (Other); Gate 21 (Unknown)
Responsible Party: Sponsor-Investigator, Ove Andersen, Research Director, MD, PhD, DMSc, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Lightel
Record Dates: First submitted 2017-08-18; First posted 2017-08-28 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Elderly Housing Residents With Frailty or Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Group 1 consists of elderly people with frailty and/or dementia living in elderly housing in Sundhedshuset, Albertslund, Denmark, and who are having CALED installed. Group 1 starts the 8 week control period and ends with the intervention consisting of 8 weeks of circadian adjusted LED-based lighting (CALED).
  Interventions: Other: 8 weeks of circadian adjusted LED-based lighting (CALED)
- Group 2 (Active Comparator): Group 2 consists of elderly people with frailty and/or dementia living in elderly housing in Sundhedshuset, Albertslund, Denmark, and who are having CALED installed. Group 2 starts with the intervention consisting of 8 weeks of circadian adjusted LED-based lighting (CALED) and ends with the 8 week control period
  Interventions: Other: 8 weeks of circadian adjusted LED-based lighting (CALED)
- Group 3. Control group (No Intervention): Group 3 consists of elderly people with frailty living in elderly housing in Sundhedshuset, Albertslund, Denmark, and who are not having CALED installed.
  This group serves as a control for:
  * Physiological or mental decline in participants during the study period
  * Seasonal variation

INTERVENTIONS:
Other: 8 weeks of circadian adjusted LED-based lighting (CALED) — The luminaires are installed before the beginning of either the control or the intervention period. During the control period (8 weeks) the luminaires have normal light. During the intervention period (8 weeks) the luminaires have CALED. Cromaviso will calibrate CALED to mimic circadian rhythm according to the latest knowledge about the light phase-response curve for elderly.
  Arms: Group 1; Group 2

SUMMARY:
Europe is undergoing a demographic change with a rapidly growing population of 65 years+. This challenges municipalities and hospitals as the ageing citizens need care and treatment due to an age-related decline in physical and mental capacity. Therefore municipalities are experiencing a growing need for sufficient and customized housing, which can support the elderly citizens in sustaining well-being and health along with preventing functional decline. Well-fare technologies, such as Circadian adjusted LED-based lighting (CALED), are suggested as a remedy for this.

To obtain proper visual sharpness and better contrast, people of older age require heightened light levels due to age-related failing vision. Furthermore, inappropriate light at night disrupts not only sleep but also the timing of the circadian rhythm, with negative consequences on cognition and emotions. Therefore CALED is being increasingly considered for use in hospitals and elderly housing because of its wide spectrum of wavelengths, good contrast and fast switching, and possibility to support a normalised circadian rhythm.

Lighting based on LED has been shown to improve the quality of sleep and to improve well-being in the elderly. However, it is not known whether CALED mimicking a normal circadian rhythm has the same benefits for elderly persons with frailty or dementia. The investigators therefore want to test the effects of CALED in elderly people with frailty and mobility disabilities and/or dementia living in elderly housing. The investigators hypothesise that CALED can improve sleep and well-being in both elderly with frailty and dementia.

DETAILED DESCRIPTION:
Due to the technical requirements, CALED will not be installed in all elderly housing facilities at Sundhedshuset, Albertslund, Denmark, limiting the number of participants receiving the intervention to 24. CALED will be installed in the residents rooms/flats and in the common areas. Residents accepting participation will comprise the following (numbers are the maximal possible): 15 elderly with frailty receiving CALED as an intervention, 9 people with dementia receiving CALED as an intervention, and 15 elderly with frailty not receiving CALED during the trial as a control group (Group 3).

The elderly receiving CALED as an intervention (15 people with frailty, 9 people with dementia) will be randomized to two groups (Group 1 and Group 2) based on equal distributions of elderly with dementia and frailty in each group and similar numbers of men and women in each group. Since the residents spend a lot of time in the same common areas where CALED is installed, the two groups are subjected to the intervention at the same time, and Group 2 therefore has a delayed start. Group 1 starts with an 8 week control period followed immediately by an 8 week intervention period. Group 2 starts with an 8 week intervention period, at the same time as Group 1, followed by and 8 week control period. Group 3 has a 16 week control period starting 4 weeks after the beginning of the control period for Group 1, and ending 4 weeks before the end of the control period for Group 2.

Timeline: Participants are included when informed consent has been obtained. CALED is installed afterwards. Randomization takes place immediately before baseline testing of Group 1, and participants are randomized by block randomization. The trial participants will be assessed at baseline, in the 4th, 8th, 12th, and 16th week, respectively. For Group 1, baseline testing takes place within two weeks prior to the beginning of the Control period. For Group 2 baseline testing takes place within two weeks prior to the beginning of the Intervention period. For Group 3 baseline testing takes place within the two weeks prior to the beginning of the Control period. See outcome measures for further details of tests.

Data collection: All data collection and assessments will be performed at "Sundhedshuset" by trained staff under the instruction and supervision of the primary investigator. Date of all assessments will be noted. Blood samples (approximately 20 ml) will be taken in "Sundhedshuset" by trained staff under the supervision of the primary investigator. Date and time of blood sampling will be documented. Blood samples will be transported to Hvidovre Hospital after collection, and plasma and serum will be stored in a biobank at -80°C until analysis.

Data management: All case report forms will be checked for errors and missing data by the assessor before being archived in a trial database and all paper-based versions will be locked in a filing cabinet in a locked room to ensure confidentiality. Data management will follow the rules of the Danish Data Protection Agency.

Power calculation: A power calculation for the Pittsburgh Sleep Quality Index (PSQI) based on a paired t-test with an alpha of 0.05, 24 pairs, a correlation of 0.8, and a standard deviation of 5.6 showed it possible to detect a minimal clinical difference of 2 with a power of 0.76. This does not account for possible drop-outs, but we expect that the inclusion of 15 control participants not exposed to CALED will increase power. Moreover, we expect that a maximum of 3 citizens will not want to participate.

We have included plasma levels of soluble urokinase plasminogen activator receptor (suPAR) as an objective and stable marker of general health status as another primary end-point. A power calculation for suPAR based on a two-sided paired t-test with an alpha of 0.05, a power of 0.8, a standard deviation of 0.5 ng/mL, and a clinical significant difference of 0.3 ng/mL (effect of healthy versus unhealthy diet is 0.35-0.55 ng/mL) gave a study population of 24 subjects. This does not account for possible drop-outs, but we expect that inclusion of 15 control participants not exposed to CALED will increase power.

Descriptive data and outcome analysis: Data will be presented as means with standard deviations, medians with inter-quartile ranges or frequencies with percentages depending on the distribution of the variable.

The primary analysis for the primary outcomes will be performed using the SAS procedure PROC MIXED (dif (intervention-control)).The difference in the PSQI scores and suPAR levels between the intervention period and the control period will be analysed using mixed models, with treatment (intervention and control) and period (period 1 and period 2) as fixed effects and the participant identification as random effect. Secondly, the models will be adjusted for baseline PSQI scores and suPAR levels, respectively. The primary analysis will follow the intention-to-treat principle using multiple imputations in case of missing outcome measures. For the secondary outcomes, similar analyses will be performed. All models will be investigated for goodness-of-fit (linearity, variance homogeneity and normal distribution of residuals) by visual inspection of plots and remodelling will be performed accordingly. All statistical tests will be performed using SAS (SAS Institute Inc., Cary, NC, USA) and p values ≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 and 2: Frail elderly (+65 years) and elderly (+50 years) with dementia, who live in the flats/rooms in Sundhedshuset, Albertslund, Denmark that have been chosen for a test installation of CALED will be invited to participate.
* Group 3: Frail elderly (+65 years) who live in the flats/rooms in Sundhedshuset, Albertslund, Denmark that have not been chosen for a test installation of CALED will be invited to participate.

Exclusion Criteria for Group 1, 2, 3:

* Terminal illness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
The average difference in Pittsburgh Sleep Quality Index (PSQI) between the end of the intervention period and the end of the control period assessed by the both participants and by staff at the nursing home. | End of intervention period (8th week assessment), end of control period (8th week assessment)
  PSQI is a measure of sleep quality consisting of 19 self-report items. Both participants and staff at the nursing home that knows the participant well evaluate the PSQI, since the participants exhibit various degrees of dementia that may affect their ability to answer the PSQI. Participants and staff indicate the amount of sleep obtained as well as factors interfering with the sleep of the participant. The subscale scores of the PSQI are summed to a total score of 0 to 21 with higher scores indicating poorer sleep quality.
  PSQI is assessed at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period. The investigators report estimates for the 8th week assessement by participants and staff, independently. Data from both the 4th and 8th week assessment will be included in the statistical model.
The average difference in plasma soluble urokinase plasminogen receptor (suPAR) between the end of the intervention period and the end of the control period. | End of intervention period (8th week assessment), end of control period (8th week assessment)
  suPAR is a stable unspecific plasma biomarker. Elevated suPAR levels are associated with morbidity and mortality, and with unhealthy lifestyle, low muscle mass, lower physical performance, and depression.
  suPAR is measured in plasma using the commercially available suPARnostic ELISA from Virogates. Plasma samples are stored in a biobank at -80°C, and measured after study completion.
  suPAR is assessed at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period. The primary analysis will follow the intention-to-treat principle (using multiple imputations). The investigators report estimates for the 8th week. Data from both the 4th and 8th week assessment will be included in the statistical model.

SECONDARY OUTCOMES:
The average difference in 24-hour mobility between the end of the intervention period and the end of the control period. | : End of intervention period (8th week assessment), end of control period (8th week assessment)
  Participants will be asked to wear an ActivPAL activity monitor (PAL Technologies Ltd, Scotland) on the thigh for one week at baseline, for one week at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period.
The average difference in Epwoth Sleepiness Scale between the end of the intervention period and the end of the control period assessed by the both participants and by staff at the nursing home. | End of intervention period (8th week assessment), end of control period (8th week assessment)
  The Epwoth Sleepiness Scale is an 8-item self-report measure in which participants indicate the likelihood of dozing off or falling asleep in eight different conditions. In addition, staff at the nursing home that knows the participant well also evaluate the Epwoth Sleepiness Scale, since the participants exhibit various degrees of dementia that may affect their ability to answer the questions. Responses are summed to a total score from 0 to 24. Higher scores indicate greater sleepiness.
  The Epwoth Sleepiness Scale is assessed at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period. The investigators report estimates for the 8th week assessment by participants and staff, independently. Data from both the 4th and 8th week assessment will be included in the statistical model.
The average difference in inflammatory biomarkers such as interleukin (IL)-6, IL-10, soluble CD14, and C reactive protein between the end of the intervention period and the end of the control period. | End of intervention period (8th week assessment), end of control period (8th week assessment)
  Inflammatory biomarkers will be measured in serum or plasma using commercially available Luminex or ELISA kits according to the manufactures instructions. Cytokines and chemokines with low systemic levels such as IL-6 will be measured with high sensitive kits to ensure detection. Samples are stored in a biobank at -80°C, and measured after study completion.
  The biomarkers are assessed at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period. The investigators report estimates for the 8th week. Data from both the 4th and 8th week assessment will be included in the statistical model.
The average difference in endocrinologic biomarkers such as insulin, glucose, cortisol, leptin and melatonin between the end of the intervention period and the end of the control period | End of intervention period (8th week assessment), end of control period (8th week assessment)
  Endocrinologic biomarkers will be measured in serum or plasma using commercially available Luminex or ELISA kits according to the manufactures instructions. Samples are stored in a biobank at -80°C, and measured after study completion.
  The biomarkers are assessed at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period. The investigators report estimates for the 8th week. Data from both the 4th and 8th week assessment will be included in the statistical model.
The average difference in the Mini Mental State Examination between the end of the intervention period and the end of the control period | End of intervention period (8th week assessment), end of control period (8th week assessment)
  The Mini Mental State Examination is an 11-item cognitive test with a maximum score of 30, with lower scores indicating more severe cognitive problems.
  The Mini Mental State Examination is conducted at baseline, in the 4th and 8th week of the intervention period, and in the 4th and 8th week of the control period. The investigators report estimates for the 8th week. Data from both the 4th and 8th week assessment will be included in the statistical model.
The average difference in the Major Depression Inventory (MDI) between the end of the intervention period and the end of the control period assessed by the both participants and by staff at the nursing home. | End of intervention period (8th week assessment), end of control period (8th week assessment)
  The MDI contains items that cover the ICD-10 symptoms of depression including DSM-IV major depression symptoms as well. The MDI contains 10 items with a maximal score of 50. In addition, staff at the nursing home that knows the participant well also evaluates the MDI, since the participants exhibit various degrees of dementia that may affect their ability to answer the questions.
  The Major Depression Inventory is conducted at baseline, in the 8th week of the intervention period, and in the 8th week of the control period. The investigators report estimates for the 8th week assessment by participants and staff independently.
The average difference in the Health related quality of life by the EuroQol (EQ-5D-3L) between the end of the intervention period and the end of the control period assessed by the both participants and by staff at the nursing home. | End of intervention period (8th week assessment), end of control period (8th week assessment)
  The three level version of the EQ-5D (EQ-5D-3L) measuring health-related quality of life by assessing aspects of physical, mental and social functioning with three response levels is used. Physical functioning is encompassed in mobility and a self-care item, social function-ing in a usual activities item, and mental functioning in an anxiety/depression item. In addition, staff at the nursing home that knows the participant well also evaluates the EQ-5D-3L, since the participants exhibit various degrees of dementia that may affect their ability to answer the questions.
  The EQ-5D-3L is conducted at baseline, in the 8th week of the intervention period, and in the 8th week of the control period. The investigators report estimates for the 8th week assessment by participants and staff independently.
The average difference in Activities of Daily living by the Barthel 20 index between the end of the intervention period and the end of the control period | End of intervention period (8th week assessment), end of control period (8th week assessment)
  The Barthel 20 Index is a performance evaluation tool assessing a person's capacity to perform 10 daily tasks without assistance and provides a summed, overall Barthel 20 Index score (0-20 points) that reflects the patient's level of independence.
  The Barthel-20 Index is assessed at baseline, in the 8th week of the intervention period, and in the 8th week of the control period.

OTHER OUTCOMES:
The average difference in mini nutritional assessment (MNA) between the end of the intervention period and the end of the control period | End of intervention period (8th week assessment), end of control period (8th week assessment)
  MNA is used to assess the nutritional status of the participants. The MNA contains 18 items, of which two are self-reported.
  MNA is assessed at baseline, in the 8th week of the intervention period, and in the 8th week of the control period.
The average difference in eyesight between the end of the intervention period and the end of the control period | End of intervention period (8th week assessment), end of control period (8th week assessment)
  We evaluate eyesight using the Snellen chart. The Snellen chart is assessed at baseline, in the 8th week of the intervention period, and in the 8th week of the control period.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, PhD, DMSc, Study Chair — Clinical Research Centre, Copenhagen University Hospital Hvidovre, Denmark
Locations (1):
- Clinical Research Centre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No